CLINICAL TRIAL: NCT00457353
Title: Phase III Comparative Study to Assess the Efficacy and Safety of Oral Rehydration Therapy (ORT) in Combination With Spores of Bacillus Clausii (Enterogermina)Versus ORT Alone, Administered for 5 Days With the Treatment of Acute Diarrhea in Children.
Brief Title: ENterogermina® (Bacillus Clausii) In the manaGeMent of diarrheA in Children
Acronym: ENIGMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENTER_L_01486
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — clausin peptide, Bacillus clausii; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Administration of oral rehydration therapy with Bacillus clausii probiotic strain (1 vial twice daily, each vial containing 2 billion spores of Bacillus clausii)
  Interventions: Drug: Bacillus Clausii
- 2 (Placebo Comparator): Administration of Oral rehydration therapy
  Interventions: Other: Oral rehydration therapy

INTERVENTIONS:
Drug: Bacillus Clausii — For 5 days
  Arms: 1
Other: Oral rehydration therapy — For 5 days
  Arms: 2

SUMMARY:
Primary:

* To demonstrate the efficacy of Enterogermina® in reducing the duration of acute diarrhea in children

Secondary:

* To evaluate the safety of Enterogermina® in acute diarrhea in Indian children

ELIGIBILITY:
Inclusion Criteria:

* Non hospitalised infants and children attending clinic/outpatients with acute diarrhea (>3 liquid or watery stools occurring in a 24-hour period) of less than 48 hours duration

Exclusion Criteria:

* History of presence of blood, pus, or mucus in stools
* Severe dehydration (World Health Organization criteria)
* Severely malnourished patients
* Treatment with antibiotics, probiotics, or prebiotics within a period of 2 weeks before enrolment
* History of conditions known to producing immunodeficiency (Acquired Immune Deficiency Syndrome, other congenital immunodeficiency syndrome, drug therapy with steroids, anticancer drugs etc)
* Known hypersensitivity to Bacillus clausii or other probiotics.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction in duration of diarrhea | Throughout the treatment period
Incidence of adverse events | Throughout the study period

SECONDARY OUTCOMES:
Mean number of stools per day | Throughout the treatment period
Effect on consistency of stools | Throughtout the treatment period
Vomiting episodes per day | Throughout the treatment period
Requirement of unscheduled intravenous transfusion | Throughout the study period
Need for hospitalization | Throughout the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Shah Pratik, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Mumbai, India